CLINICAL TRIAL: NCT01317173
Title: The Impact of FGF23 and Klotho on Progression of Chronic Kidney Disease
Brief Title: Factors Related to the Progression of Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Alper AZAK, Ankara Education and Research Hospital
Other Study IDs: NEPH001
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease progression; FGF 23; Klotho
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Progressive disease: Serum creatinin level rise more than 2 times
- Non-progressive disease: Serum creatinin level rise less than 2 times

SUMMARY:
Chronic kidney disease is a progressive disorder that has been influenced with many factors. Most of the patients has altered Ca P metabolism and these dis orders are the contributing factors of the disease progression. It has been recently documented that FGF23 and Klotho are the key factors of PTH secretion Ca-P metabolism. This study aimed to evaluate the impact of Klotho and FGF23 on the progression of stage 3-4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic chronic kidney disease

Exclusion Criteria:

* Presence of DM
* Actively using calcium based phosphorus binder of vitamin D

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-diabetic chronic kidney disease between the ages of 18 and 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Progression of kidney disease | continuous measurement of kidney functions 3 monthly for two years or until the outcome reached
  Doubling of creatinin, requirement of renal replacement therapy

SECONDARY OUTCOMES:
Evaluation of Ca P metabolism | 3 monthly for two years or until the outcome reached
  Determination of Ca-P metabolism disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Education and Research Hospital, Ankara, Turkey (Türkiye)